CLINICAL TRIAL: NCT06256237
Title: Neoadjuvant Therapy With Toripalimab and JS004 Combined With Etoposide and Platinum Chemotherapy for Limited-stage Small Cell Lung Cancer : A Single-arm, Phase 2 Trial
Brief Title: Neoadjuvant Therapy With Toripalimab and JS004 Combined With Etoposide and Platinum Chemotherapy for Limited-stage Small Cell Lung Cancer : A Phase 2 Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Peng Zhang, Director, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LungMate-023
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Limited Stage Small Cell Lung Cancer
Keywords: small cell lung cancer; Toripalimab; JS004; Limited Stage
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — toripalimab; Surgical Procedures, Operative; Etoposide; Platinum

STUDY DESIGN:
Intervention Model Description: All enrolled patients received toripalimab and JS004 Combined With etoposide and platinum Chemotherapy.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant Therapy With Toripalimab and JS004 Combined With Etoposide and Platinum Chemotherapy (Experimental): In this arm, 30 patients with limited-stage small cell lung cancer will receive 4 circles of neoadjuvant toripalimab and JS004 combined with etoposide and platinum chemotherapy. And those resectable after neoadjuvant therapy will be treated with surgery. Postoperative patients receive two cycles of toripalimab and JS004 combined with etoposide and platinum chemotherapy. then patients received maintenance treatment with toripalimab and JS004 until the disease progressed.
  Interventions: Drug: JS004; Drug: Toripalimab; Procedure: surgery; Drug: Etoposide; Drug: Platinum

INTERVENTIONS:
Drug: JS004 — Specified dose on specified days.
  Other Names: tifcemalimab
Drug: Toripalimab — Specified dose on specified days.
Procedure: surgery — Patients with resectable tumors after neoadjuvant therapy will be treated with surgery.
Drug: Etoposide — Specified dose on specified days.
Drug: Platinum — Specified dose on specified days.

SUMMARY:
For limited-stage small cell lung cancer (SCLC), neoadjuvant chemotherapy plus PD-1 antibody is recommended. However, most patients cannot achieve a complete pathological response (CPR). A new immunotherapeutic strategy is needed to achieve a higher CPR rate. JS004 is a new antibody targeting B and T lymphocyte attenuator (BTLA), which restrains immune cells' function and leads to immune escape of tumor cells. The combination of PD-1 and BTLA antibodies has shown a good therapeutic effect in solid tumors. This trial aims to investigate the efficacy and safety of the therapeutic regimen of toripalimab and JS004 plus etoposide and platinum Chemotherapy in limited-stage SCLC.

ELIGIBILITY:
Inclusion Criteria:

1. The patient shall sign the Informed Consent Form.
2. Aged 18 ≥ years.
3. Histological or cytological diagnosis of SCLC by needle biopsy, and limited stage confirmed by imageological examinations (CT, PET-CT or EBUS).
4. Eastern Cooperative Oncology Group (ECOG) performance-status score of 0 or 1.
5. Life expectancy is at least 12 weeks.
6. At least 1 measurable lesion according to RECIST 1.1.
7. Patients with good function of other main organs (liver, kidney, blood system, etc.)
8. Without systematic metastasis (including M1a, M1b and M1c);
9. Expected to be completely resected
10. Patients with lung function can tolerate surgery
11. Fertile female patients must voluntarily use effective contraceptives not less than 120 days after chemotherapy or the last dose of toripalimab (whichever is later) during the study period, and urine or serum pregnancy test results within 7 days prior to enrollment are negative.
12. Unsterilized male patients must voluntarily use effective contraception during the study period not less than 120 days after chemotherapy or the last dose of toripalimab (whichever is later).

Exclusion Criteria:

1. Participants who have received any systemic anti-cancer treatment for thymic epithelial tumor, including surgical treatment, local radiotherapy, cytotoxic drug treatment, targeted drug treatment and experimental treatment;
2. Patients with a malignancy other than SCLC within five years prior to the start of this trial;
3. Participants with any unstable systemic disease (including active infection, uncontrolled hypertension), unstable angina pectoris, angina pectoris starting in the last three months, congestive heart failure (>= NYHA) Grade II), myocardial infarction (6 months before admission), severe arrhythmia requiring drug treatment, liver, kidney or metabolic diseases;
4. With activate or suspectable autoimmune disease, or autoimmune paracancer syndrome requiring systemic treatment;
5. Participants who are allergic to the test drug or any auxiliary materials;
6. Participants with Interstitial lung disease currently;
7. Participants with active hepatitis B, hepatitis C or HIV;
8. Pregnant or lactating women;
9. Any malabsorption;
10. Participants suffering from nervous system diseases or mental diseases that cannot cooperate
11. Other factors that researchers think it is not suitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2032-01-31 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response (PCR) rate | Up to 30 months
  PCR rate is defined as the proportion of participants who have achieved pathologic complete response (on routine hematoxylin and eosin staining, no tumor cell can be found in tumor bed or lymph node) in all participants.

SECONDARY OUTCOMES:
Objective response rate (ORR) | up to 30 months
  ORR is defined according to the RECIST v1.1 criteria.
Major pathologic response (MPR) rate | Up to 30 months
  MPR rate is defined as the proportion of participants who have achieved major pathologic response (on routine hematoxylin and eosin staining, tumors with no more than 10% viable tumor cells) in all participants.
Treatment-related adverse event (TRAE) | Up to 30 months
  TRAE is defined and classified according to NCI-CTCAE v5.0 in all participants.
Event-free survival (EFS) | up to 60 months
  Event-free survival (EFS) is defined as the length of time (months) from randomization to any of the following events: any progression of disease precluding surgery, progression or recurrence disease based on response evaluation criteria in solid tumors (RECIST) 1.1 after surgery, or death due to any cause. Participants who don't undergo surgery for reason other than progression will be considered to have an event at progression or death. Progression is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Overall survival (OS) | up to 60 months
  It is defined as the time (months) from enrollment to death of participant due to any cause. In the case of a patient who still survives at the time of analysis, the date of last contact will be taken as the censoring date.
EORTC-QLQ-C30 scale | up to 5 months
  The assessment is made according to the Quality of Life Scale for Lung Cancer Patients (EORTC-QLQ-C30, Version 3). EORTC's QLQ-C30 (V3.0) is a core scale for lung cancer patients, with a total of 30 items. Among them, Item 29 and 30 are divided into seven grades, which are assigned with 1 to 7 scores according to the answer options. The other items are divided into 4 grades: Not at All, A Little, Quite a Bit, and Very Much, assigned with 1 to 4 scores respectively. The higher score, the worse quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided
The researchers will consider whether IPD is available to other researchers only after the paper is published.